CLINICAL TRIAL: NCT02432092
Title: Pediatric Cardiomyopathy Mutation Analysis
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Stephanie Ware, Professor of Pediatrics and Medical and Molecular Genetics, Indiana University
Other Study IDs: 1403919054
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Cardiomyopathies; Dilated Cardiomyopathy; Hypertrophic Cardiomyopathy; Restrictive Cardiomyopathy; Arrhythmogenic Right Ventricular Cardiomyopathy; Left Ventricular Non-compaction Cardiomyopathy
Keywords: Cardiomegaly; Cardiovascular Diseases; Heart Diseases; Systolic dysfunction; Diastolic dysfunction; Ventricular hypertrophy; Heart failure
MeSH Terms: conditions — Cardiomyopathies; Cardiomyopathy, Dilated; Cardiomyopathy, Hypertrophic; Cardiomyopathy, Restrictive; Arrhythmogenic Right Ventricular Dysplasia; Cardiomegaly; Cardiovascular Diseases; Heart Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, Saliva, Tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Affected: participants with cardiomyopathy
- Family Members of affected: Family members of participants with cardiomyopathy (can be affected or unaffected)

SUMMARY:
The goal of this protocol is to obtain information from individuals with cardiomyopathy and from their families in order to elucidate the molecular genetics of this disorder. This will provide the basis for future genetic counseling as well as contribute to elucidating the biology of normal and abnormal cardiac function.

DETAILED DESCRIPTION:
Cardiomyopathy is a genetically heterogeneous heart muscle disorder that results in ventricular dysfunction. While significant progress has been made in identifying the genetic basis of cardiomyopathy in adults, molecular diagnosis in children has proven more challenging and current algorithms do not incorporate mutation analysis in the clinical protocol. However, recent studies indicate that cardiomyopathy outcomes in children are origin specific, highlighting the importance of precise diagnosis. The goal of this study is to identify the genetic causes of pediatric cardiomyopathy. Rapid, comprehensive and cost-effective detection of genetic causes of cardiomyopathy will aid management and development of novel treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with cardiomyopathy
* Family members of subjects with cardiomyopathy

Exclusion Criteria:

* Subjects without cardiomyopathy
* Family members of subjects without cardiomyopathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Families affected by cardiomyopathy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-04; Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Elucidate the molecular genetics of cardiomyopathy | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Ware, MD, PhD, Principal Investigator — IU School of Medicine
Locations (1):
- IU School of Medicine, Indianapolis, Indiana, United States